CLINICAL TRIAL: NCT03902834
Title: Move for Surgery (MFS): Evaluating the Use of Wearable Technology for Preconditioning Before Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Wael Hanna, Assistant Professor of Surgery, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BFCRS-333417
Record Dates: First submitted 2018-01-30; First posted 2019-04-04 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Preconditioning; Lung Cancer, Nonsmall Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Other: Fitbit

INTERVENTIONS:
Other: Fitbit — Use the wearable technology (Fitbit) and proven behavioural change techniques to precondition patients prior to lung cancer surgery
  Other Names: Wearable Technology

SUMMARY:
Wearable technology is increasingly being used to promote healthy behaviour. In this study, the investigators propose the development and evaluation of Move for Surgery, which utilizes a wearable activity bracelet (Fitbit) and proven behavioural change techniques, for preconditioning of patients prior to lung cancer surgery. The primary outcome of this study will be compliance with Move for Surgery, as a surrogate measure for feasibility. Secondary outcomes, including accrual rates, perioperative pulmonary complications, cost per patient, and patient satisfaction, will also be collected. The investigators have partnered with the Canadian Partnership Against Cancer (CPAC) and Lung Cancer Canada (LCC) to develop Move for Surgery. The ultimate goal of this preliminary study is to lay the groundwork for a subsequent comparative trial to evaluate the impact of Move for Surgery on postoperative complications in the thoracic surgery population.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants include patients with NSCLC set to undergo pulmonary resection.

Exclusion Criteria:

* There will be no exclusion based on functional status in this feasibility study; rather, a subsequent analysis of participant demographics will be performed to inform future phases of this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
The feasibility of Move for Surgery, as measured by a rate of compliance of >70% until program completion. | 12 months
  The feasibility of Move for Surgery, as measured by a rate of compliance of >70% until program completion.

SECONDARY OUTCOMES:
Rate of accrual | 12 months
  Rate of accrual
Perioperative patient complications | 12 months
  Perioperative patient complications
Cost per patient | 12 months
  Cost per patient
Patient-reported health-related quality of life | 12 months
  EuroQol-5Dimensions-5Levels (EQ-5D-5L)
Patient-reported health-related physical activity | 12 months
  International Physical Activity Questionnaire - Short Form (IPAQ-SF)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No